CLINICAL TRIAL: NCT01931098
Title: A Phase II Trial of Oral Pazopanib Plus Oral Topotecan Metronomic Antiangiogenic Therapy for Recurrent Glioblastoma Multiforme (A)Without Prior Bevacizumab Exposure and (B) After Failing Prior Bevacizumab
Brief Title: Oral Pazopanib Plus Oral Topotecan Metronomic Antiangiogenic Therapy for Recurrent Glioblastoma Multiforme (A) Without Prior Bevacizumab Exposure and (B) After Failing Prior Bevacizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Camphausen, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160034; 16-C-0034
Record Dates: First submitted 2013-08-23; First posted 2013-08-29 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Gliosarcoma; Brain Neoplasms; Central Nervous System Neoplasms
Keywords: Brain Tumors
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms; Central Nervous System Neoplasms | interventions — Topotecan; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glioblastoma or Gliosarcoma With No Prior Bevacizumab Exposure (Experimental): Topotecan .25 mg and pazopanib 600 mg are administered orally daily until progression, up to one year.
  Interventions: Drug: topotecan; Drug: pazopanib
- Glioblastoma or Gliosarcoma With Prior Bevacizumab Exposure (Experimental): Topotecan .25 mg and pazopanib 600 mg are administered orally daily until progression, up to one year.
  Interventions: Drug: topotecan; Drug: pazopanib

INTERVENTIONS:
Drug: topotecan — Taken .25 mg orally, daily continuous until progression up to one year.
  Other Names: Hycamtin
Drug: pazopanib — 600 mg orally, daily until progression, up to one year.
  Other Names: Votrient

SUMMARY:
Background:

Glioblastoma is the most common and most aggressive type of malignant brain tumor. The drug pazopanib is used to treat people with a type of kidney cancer. Topotecan is used to treat lung cancer. Both topotecan and pazopanib have individually been used to treat patients with glioblastoma and some anti-tumor activity has been found. Researchers want to see if these two drugs together may be able to help people with glioblastoma.

Objectives:

To learn if pazopanib with topotecan can help control glioblastoma. Also, to study the safety of this drug combination.

Eligibility:

Adults at least 18 years old whose glioblastoma has returned after treatment.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Brain computed tomography (CT) or magnetic resonance imaging (MRI) For these, participants lay in a machine that takes pictures.

Chest CT scan or x-ray

Heart electrocardiogram (EKG)

A questionnaire about quality of life

Participants will be assigned to a study group.

Participants will take the study drugs for 28-day cycles for up to 1 year. They will take capsules of topotecan by mouth once every day. They will take tablets of pazopanib by mouth once every day.

Participants will write in a diary the times they take the study drugs.

Participants will have several study visits during each cycle. These may include

Blood pressure measurement

Blood and urine tests

EKG

Physical exam and/or neurological exam

Brain MRI or CT scan to check the status of the disease

A symptom questionnaire

At the end of treatment, participants will have a physical exam. They may have blood drawn.

Participants will have follow-up calls once every 3 months to check.

DETAILED DESCRIPTION:
Background

* Glioblastoma (GBM) is the most common primary brain tumor. With optimal treatment,consisting of focal radiotherapy with concurrent chemotherapy, followed by adjuvant chemotherapy, median survival is 14.6 months. Most patients have evidence of tumor progression within one year of diagnosis despite treatment. At progression, treatment options are limited and mostly ineffective.
* Recently, bevacizumab was approved for recurrent GBM patients who fail bevacizumab indicate a short survival, on the order of 10 weeks, an approximate PFS 3 and 6 months of 0%.
* Pazopanib is an oral angiogenesis inhibitor targeting vascular endothelial growth factor (VEGFR), Platelet-derived growth factor receptors (PDGFR), and c-Kit, and was recently Food and Drug Administration (FDA) approved for advanced renal cell carcinoma.
* Topotecan is an orally bioavailable topoisomerase I and Hypoxia-inducible factor 1 (HIF-1) alpha inhibitor with reasonably high central nervous system (CNS)/cerebrospinal fluid (CSF) penetration
* Recent pre-clinical reports have begun to argue for the clinical testing of metronomic chemotherapy administration in various cancers. The theory of improved activity of Pazopanib + Topotecan administered metronomically is based on targeting tumor vasculature (both existing capillary endothelial cells and circulating bone marrow derived endothelial cell precursors), immune modulation, as well as tumor cell HIF-1 alpha inhibition, and the induction of Deoxyribonucleic acid (DNA) damage. Further support for the combination comes from recent data tying drug-induced VEGF inhibition to the induction of HIF-1 alpha activity in GBM suggesting possible synergy between Pazopanib and Topotecan
* The combination of Topotecan and Pazopanib has been directly demonstrated as active in

animal models

Objectives

* 6 month progression free survival rate for recurrent glioblastoma (rGBM) patients with no prior bevacizumab exposure treated with pazopanib and topotecan (Group A).
* 3 month progression free survival rate for rGBM patients with prior bevacizumab exposure treated with pazopanib and topotecan (Group B).

Eligibility

* Histologically proven intracranial glioblastoma multiforme (GBM) or gliosarcoma (GS) with evidence of progression on MRI or CT scan.
* Patient must have failed prior chemoradiation with temozolomide and any other therapies except Bevacizumab (BEV) (group A), or must have failed primary chemoradiation and a BEVincorporating treatment (group B).
* Patients must be greater than 12 weeks following completion of chemoradiation.

  * Archived tumor tissue must be available for confirmation of the diagnosis
  * Patients must be > 18 years old.
  * Patients must have a Karnofsky performance status of > 60.
  * Patients must have adequate organ function.
  * No pregnancy or lactation.
  * Patients must not have any significant medical illnesses that in the investigators opinion cannot be adequately controlled with appropriate therapy or would compromise the patients ability to tolerate this therapy.
  * No history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are eligible.
  * No clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, or the absorption of the medications.
  * No prior major surgery or trauma within 28 days and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
  * No evidence of active bleeding or bleeding diathesis.
  * No known endobronchial lesions and/or lesions infiltrating major pulmonary vessels.
  * No serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subjects safety, provision of informed consent, or compliance to study procedures.
  * No ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity, except alopecia.
  * No ongoing use of enzyme-inducing anti-epileptic agents (EIAEDs), unless 2 week washout has elapsed form last dose of EIAED.
  * No known hypersensitivity to pazopanib or topotecan or to their excipients.
  * No total daily dose of dexamethasone greater than 16 mg/day.
  * No prior therapy with topotecan, pazopanib, or related drugs such as tyrosine kinase inhibitors, VEGF inhibitors (except bevacizumab). Prior treatment with Tyrosine kinase inhibitors (TKIs) that do not impact VEGFR -1, -2, or -3, Platelet Derived Growth Factor Receptor Alpha (PDGFRa) Platelet Derived Growth Factor Receptor Beta (-b) of cKIT could be allowed.

Design

This is a 2 arm phase II trial of the combination of topotecan and pazopanib in patients with recurrent GBM or GS. Patients will be enrolled into one of the following groups: (A) Glioblastoma or gliosarcoma with no prior bevacizumab exposure: (B) Glioblastoma or

gliosarcoma with prior bevacizumab exposure. Topotecan and pazopanib are administered orally daily. The primary efficacy endpoint is progression free survival (PFS) at six months from patient registration for bevacizumab na(SqrRoot) ve patients and progression free survival (PFS) at 3 months for patients with prior bevacizumab treatment.

ELIGIBILITY:
* General Inclusion Criteria
* Patients with histologically proven intracranial glioblastoma multiforme (GBM) or gliosarcoma (GS). Patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a GBM or GS is made. Patients must have evidence of progression of the GBM or GS on magnetic resonance imaging (MRI) or computed tomography (CT) scan. Patient must have failed prior chemoradiation with temozolomide and any other therapies except BEV (group A), or must have failed primary chemoradiation and a BEV-incorporating treatment (group B).
* Patients may have had treatment for no more than 2 prior relapses. Relapse is defined as progression following initial therapy (i.e. radiation+/- chemo if that was used as initial therapy). The intent therefore is that patients had no more than 3 prior therapies

(initial and treatment for 2 relapses). If the patient had a surgical resection for relapsed disease and no anti-cancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered as 1 relapse.

For patients who had prior therapy for a low-grade glioma, the surgical diagnosis of a high-grade glioma will be considered the first relapse.

* Patients must be greater than 12 weeks following completion of chemoradiation or any additional radiation to reduce the chance of pseudoprogression.
* Measurable disease is required unless patient is post-operative and in that case patient can have no evidence of disease.
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study.
* Archived tumor tissue must be available for all subjects for confirmation of the diagnosis before or during treatment. Samples must be provided within 4 weeks of enrollment.
* Patients must be greater than or equal to 18 years old.
* Patients must have a Karnofsky performance status of greater than or equal to 60.
* At the time of registration: Patients must have recovered from the toxic effects of prior therapy: greater than or equal to 28 days from any investigational agent, greater than or equal to 28 days from prior cytotoxic therapy, greater than or equal to 14 days from vincristine, greater than or equal to 42 days from nitrosoureas, greater than or equal to 21 days from procarbazine administration, >21 days from bevacizumab administration and greater than or equal to 7 days for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of noncytotoxic agents should be directed to Academic Principal Investigator (PI).
* Patients must have adequate organ function:

  * Bone marrow function (White blood cell (WBC) greater than or equal to 3,000/microl, absolute neutrophil count (ANC) greater than or equal to 1,500/mm^3, platelet count of greater than or equal to 100,000/mm^3, and hemoglobin greater than or equal to 10 gm/dl).

    ---Eligibility level for hemoglobin may be reached by transfusion.
  * Liver function (alanine amino transferase (ALT) and aspartate aminotransferase (AST) < 2.5 X upper limit of normal (ULN), and total bilirubin < 1.5 X ULN), prothrombin time (PT) or international normalized ratio (INR), and activated partial thromboplastin time (aPTT) less than or equal to 1.2 X ULN.

    * Concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN (upper limit of normal) are not permitted.
    * Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation.
  * Renal function (creatinine less than or equal to 1.5 mg/dL (133 micromol/L), or if > 1.5 mg/dL, calculated creatinine clearance greater than or equal to 50 cc/min), and urine protein to creatinine ratio of < 1 prior to registration.
* Patients must have shown unequivocal radiographic evidence for tumor progression by MRI or CT scan as defined by Section 6.4.1.4.5. A scan should be performed within 14 days prior to registration and on a steroid dose that has been stable or decreasing for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline MR/CT is required. The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement.
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

  --They have recovered from the effects of surgery and be > 28 days from surgery.
* Residual disease following resection of recurrent GBM or GS is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a CT/ MRI should be done no later than 96 hours in the immediate post-operative period or at least 4 weeks post-operatively, within 14 days prior to registration. If the 96-hour scan is more than 14 days before registration, the scan needs to be repeated. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required on a stable steroid dosage for at least 5 days.
* Patients must have failed prior radiation therapy and must have an interval of greater than or equal to 12 weeks from the completion of radiation therapy to study entry.
* Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based upon either positron emission tomography (PET) or Thallium scanning, MR spectroscopy or surgical/pathological documentation of disease.
* A female is eligible to enter and participate in this study if she is of:

  * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:

    * A hysterectomy
    * A bilateral oophorectomy (ovariectomy)
    * A bilateral tubal ligation
    * Is post-menopausal
    * Subjects not using hormone replacement therapy (HRT) must have experienced in questionable cases, have a follicle stimulating hormone (FSH) value >40 mIU/mL and an estradiol value < 40pg/mL (<140 pmol/L).
    * Subjects using HRT must have experienced total cessation of menses for >= 1year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT
  * Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. Novartis acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:

    * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product. Oral contraceptive, either combined or progestogen alone.
    * Injectable progestogen.
    * Implants of levonorgestrel.
    * Estrogenic vaginal ring.
    * Percutaneous contraceptive patches.
    * Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year.
    * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject.
    * Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository).
    * Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

General Exclusion Criteria

* Patients must not have any significant medical illnesses that in the investigators opinion cannot be adequately controlled with appropriate therapy or would compromise the patients ability to tolerate this therapy.
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

  * Active peptic ulcer disease.
  * Known intraluminal metastatic lesion/s with risk of bleeding.
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation.
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment.
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

  * Malabsorption syndrome
  * Major resection of the stomach or small bowel.
  * Presence of uncontrolled infection.
  * Corrected QT interval (QTc) > 480 msecs using Bazett's formula. Bazett's Formula: QTc (Bazett)=QT/RR
* History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA), see appendix 13.7
  * Poorly controlled hypertension [defined as systolic blood pressure (SBP) of greater than or equal to 140 mmHg or diastolic blood pressure (DBP) of less than or equal to 90mmHg]. Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. BP must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP/DBP values from each BP assessment must be less than or equal to 140/90 mmHg in order for a subject to be eligible for the study.
  * History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anticoagulating

agents for at least 6 weeks are eligible.

* Prior major surgery or trauma within 28 days and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* Hemoptysis in excess of 2.5 mL (or one half teaspoon) within 8 weeks of first dose of study drug.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subjects safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of inducers and inhibitors of Cytochrome P450 (CYP450) listed in Appendix 13.4 and breast cancer resistance protein (BCRP) and P-glycoprotein (PgP) inducers and inhibitors for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study. (CYP3A4 substrates can be administered, but investigators will need to be aware of possible increased or decreased effectiveness of the non-study drug and this should be recorded in concomitant medications. Dexamethasone is acceptable although listed as a CYP3A4 inducers/inhibitors as long as the dose is 16 mg/day or lesser.
* Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity, except alopecia.
* Ongoing use of enzyme-inducing anti-epileptic agents (EIAEDs), unless 2 week washout has elapsed form last dose of EIAED.
* Patients must not have any significant medical illnesses that in the investigators opinion cannot be adequately controlled with appropriate therapy or would compromise the patients ability to tolerate this therapy.
* Patients with a known hypersensitivity to pazopanib or topotecan or to their excipients.
* Patients on total daily dose of dexamethasone greater than 16 mg/day.
* Patients must not have received prior therapy with topotecan, pazopanib, or related drugs such as tyrosine kinase inhibitors, VEGF inhibitors (except bevacizumab). Prior treatment with TKIs that do not impact VEGFR -1, -2, or -3, Platelet Derived Growth Factor Receptor Alpha (PDGFRa) Platelet Derived Growth Factor Receptor Beta (-b) of cKIT could be allowed.
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macdonald D, Cairncross G, Stewart D, Forsyth P, Sawka C, Wainman N, Eisenhauer E. Phase II study of topotecan in patients with recurrent malignant glioma. National Clinical Institute of Canada Clinical Trials Group. Ann Oncol. 1996 Feb;7(2):205-7. doi: 10.1093/oxfordjournals.annonc.a010550. PMID 8777179
- [Background] Armstrong TS, Mendoza T, Gning I, Coco C, Cohen MZ, Eriksen L, Hsu MA, Gilbert MR, Cleeland C. Validation of the M.D. Anderson Symptom Inventory Brain Tumor Module (MDASI-BT). J Neurooncol. 2006 Oct;80(1):27-35. doi: 10.1007/s11060-006-9135-z. Epub 2006 Apr 6. PMID 16598415
- [Background] Vredenburgh JJ, Desjardins A, Herndon JE 2nd, Marcello J, Reardon DA, Quinn JA, Rich JN, Sathornsumetee S, Gururangan S, Sampson J, Wagner M, Bailey L, Bigner DD, Friedman AH, Friedman HS. Bevacizumab plus irinotecan in recurrent glioblastoma multiforme. J Clin Oncol. 2007 Oct 20;25(30):4722-9. doi: 10.1200/JCO.2007.12.2440. PMID 17947719
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0034.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Glioblastoma or Gliosarcoma With No Prior Bevacizumab Exposure; Glioblastoma or Gliosarcoma With Prior Bevacizumab Exposure: Topotecan and pazopanib are administered orally daily.
  topotecan: Taken .25 mg orally, daily continuous until progression up to one year.
  pazopanib: 600 mg orally, daily until progression, up to one year.
Period: Overall Study
Arm/Group | Glioblastoma or Gliosarcoma With No Prior Bevacizumab Exposure | Glioblastoma or Gliosarcoma With Prior Bevacizumab Exposure
Started | 9 | 26
Completed | 9 | 22
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Enrolled in different protocol | 0 | 1
Not completed — Unable to begin trmt:active infection | 0 | 1
Not completed — Refused further treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glioblastoma or Gliosarcoma With No Prior Bevacizumab Exposure | Glioblastoma or Gliosarcoma With Prior Bevacizumab Exposure | Total
Number analyzed (Participants) | 9 | 26 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 22 | 29
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (9.51) | 50.81 (13.26) | 51.79 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 4 | 15 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 26 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 26 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 26 | 35

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients That Have Progressive Survival (PFS) at Six Months From Patient Registration for Bevacizumab Naive Patients and PFS at 3 Months for Patients With Prior Bevacizumab Treatment
Description: PFS was evaluated using the Kaplan-Meier product-limit survival curve methodology. For participants with no prior bevacizumab exposure, PFS is defined as 2 or more participants who are progression free at 6 months. For participants with prior bevacizumab exposure, PFS is defined as 1 or more participants who are progression free at 3 months. Progression is a 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) or clear worsening of evaluable disease or the appearance of any new lesions.
Time Frame: six months from patient registration for bevacizumab naive patients, and 3 months from patient registration for patients with prior bevacizumab treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Glioblastoma or Gliosarcoma With No Prior Bevacizumab Exposure | Glioblastoma or Gliosarcoma With Prior Bevacizumab Exposure
Number analyzed (Participants) | 9 | 26
proportion of participants
  3 months | 0.44 [0.14 to 0.72] | 0.18 [0.06 to 0.36]
  6 months | 0.11 [0.01 to 0.39] | 0 [0 to 0]

2. Secondary Outcome: Overall Survival
Description: OS was evaluated using the Kaplan-Meier product-limit survival curve methodology and is defined as the time from date of registration to date of death due to any cause.
Time Frame: From date of registration to date of death due to any cause, up to 5 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Glioblastoma or Gliosarcoma With No Prior Bevacizumab Exposure | Glioblastoma or Gliosarcoma With Prior Bevacizumab Exposure
Number analyzed (Participants) | 9 | 26
Months | 7.1 [2.9 to 8.2] | 6.3 [2.8 to 9.1]

3. Secondary Outcome: Mean Symptom Severity Score Between Responders and Non-responders at Baseline and by Cycle
Description: Responders and Non-Responders symptom presence and severity were assessed by the M.D. Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) questionnaire using an scale of (0-10); 0 being not present and 10 being the worst, and Responders were defined as patients with stable disease (SD) and partial response (PR) as their best response, and Non-responders were defined as patients with disease progression (PD) as their best response. Partial response is greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesion. Progressive disease is a 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease). And stable disease does not qualify for complete response, partial response or progression.
Time Frame: Baseline, and Cycles 1-6
Population: One participant in the second Arm/Group did not have a best response recorded and was excluded from questions involving responders and non-responders.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Glioblastoma or Gliosarcoma With No Prior Bevacizumab Exposure: Participants received imaging and corresponding MDSAI-BT at baseline and even-numbered cycles.
- Glioblastoma or Gliosarcoma With Prior Bevacizumab Exposure: Participants received imaging and corresponding MDSAI-BT at baseline and cycle 1 thru cycle 3, and subsequent odd-numbered cycles.
Arm/Group | Glioblastoma or Gliosarcoma With No Prior Bevacizumab Exposure | Glioblastoma or Gliosarcoma With Prior Bevacizumab Exposure
Number analyzed (Participants) | 9 | 25
scores on a scale
  Responders - baseline: number analyzed (Participants) | 6 | 12
  Responders - baseline | 1.1 (0.4) | 1.9 (1.3)
  Responders - Cycle 1: number analyzed (Participants) | 0 | 10
  Responders - Cycle 1 |  | 2.3 (1.4)
  Responders - Cycle 2: number analyzed (Participants) | 3 | 8
  Responders - Cycle 2 | 0.8 (0.4) | 3.5 (2.5)
  Responders - Cycle 3: number analyzed (Participants) | 0 | 4
  Responders - Cycle 3 |  | 2.9 (3.4)
  Responders - Cycle 4: number analyzed (Participants) | 4 | 0
  Responders - Cycle 4 | 2.0 (1.7) |
  Responders - Cycle 5: number analyzed (Participants) | 0 | 1
  Responders - Cycle 5 |  | 1.5
  Responders - Cycle 6: number analyzed (Participants) | 2 | 0
  Responders - Cycle 6 | 2.1 (2.0) |
  Non-Responders - baseline: number analyzed (Participants) | 3 | 8
  Non-Responders - baseline | 1.6 (0.7) | 2.8 (2.1)
  Non-Responders - Cycle 1: number analyzed (Participants) | 0 | 5
  Non-Responders - Cycle 1 |  | 3.0 (1.9)
  Non-Responders - Cycle 2: number analyzed (Participants) | 1 | 0
  Non-Responders - Cycle 2 | 3.0 |
  Overall Responders and Non-Responders - baseline: number analyzed (Participants) | 9 | 21
  Overall Responders and Non-Responders - baseline | 1.3 (0.5) | 2.4 (1.7)
  Overall Responders and Non-Responders - Cycle 1: number analyzed (Participants) | 0 | 15
  Overall Responders and Non-Responders - Cycle 1 |  | 2.5 (1.5)
  Overall Responders and Non-Responders - Cycle 2: number analyzed (Participants) | 4 | 8
  Overall Responders and Non-Responders - Cycle 2 | 1.4 (1.2) | 3.5 (2.5)
  Overall Responders and Non-Responders - Cycle 3: number analyzed (Participants) | 0 | 4
  Overall Responders and Non-Responders - Cycle 3 |  | 2.9 (3.4)
  Overall Responders and Non-Responders - Cycle 4: number analyzed (Participants) | 4 | 1
  Overall Responders and Non-Responders - Cycle 4 | 2.0 (1.7) | 1.5
  Overall Responders and Non-Responders - Cycle 5: number analyzed (Participants) | 0 | 0
  Overall Responders and Non-Responders - Cycle 6: number analyzed (Participants) | 2 | 0
  Overall Responders and Non-Responders - Cycle 6 | 2.1 (2.0) |

4. Secondary Outcome: Mean Symptom Interference Score Between Responders and Non-responders at Baseline and by Cycle
Description: Responders and Non-Responders symptom interference was assessed by the M.D. Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) questionnaire that determined how much general activity, mood, work inside and outside the home, relations with other people, walking and enjoying life interfered with a participant's life rated on an scale (0-10); 0 being not present and 10 being the worst. Responders were defined as patients with stable disease (SD) and partial response (PR) as their best response, and Non-responders were defined as patients with disease progression (PD) as their best response. Partial response is greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesion. Progressive disease is a 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease). And stable disease does not qualify for complete response, partial response or progression.
Time Frame: Baseline, and Cycles 1-6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Glioblastoma or Gliosarcoma With No Prior Bevacizumab Exposure | Glioblastoma or Gliosarcoma With Prior Bevacizumab Exposure
Number analyzed (Participants) | 9 | 25
scores on a scale
  Responders - baseline: number analyzed (Participants) | 6 | 12
  Responders - baseline | 2.1 (1.2) | 3.6 (2.9)
  Responders - Cycle 1: number analyzed (Participants) | 0 | 10
  Responders - Cycle 1 |  | 3.7 (2.5)
  Responders - Cycle 2: number analyzed (Participants) | 3 | 8
  Responders - Cycle 2 | 1.4 (0.4) | 6.0 (3.2)
  Responders - Cycle 3: number analyzed (Participants) | 0 | 4
  Responders - Cycle 3 |  | 4.2 (4.0)
  Responders - Cycle 4: number analyzed (Participants) | 4 | 0
  Responders - Cycle 4 | 3.2 (2.0) |
  Responders - Cycle 5: number analyzed (Participants) | 0 | 1
  Responders - Cycle 5 |  | 0.2
  Responders - Cycle 6: number analyzed (Participants) | 2 | 0
  Responders - Cycle 6 | 2.7 (0.9) |
  Non-Responders - baseline: number analyzed (Participants) | 3 | 8
  Non-Responders - baseline | 1.7 (1.2) | 3.9 (3.2)
  Non-Responders - Cycle 1: number analyzed (Participants) | 0 | 5
  Non-Responders - Cycle 1 |  | 4.8 (3.8)
  Non-Responders - Cycle 2: number analyzed (Participants) | 1 | 0
  Non-Responders - Cycle 2 | 3.0 |
  Overall Responders and Non-Responders - baseline: number analyzed (Participants) | 9 | 21
  Overall Responders and Non-Responders - baseline | 2.0 (1.2) | 3.8 (2.9)
  Overall Responders and Non-Responders - Cycle 1: number analyzed (Participants) | 0 | 15
  Overall Responders and Non-Responders - Cycle 1 |  | 4.0 (2.9)
  Overall Responders and Non-Responders - Cycle 2: number analyzed (Participants) | 4 | 8
  Overall Responders and Non-Responders - Cycle 2 | 1.8 (0.9) | 6.0 (3.2)
  Overall Responders and Non-Responders - Cycle 3: number analyzed (Participants) | 0 | 4
  Overall Responders and Non-Responders - Cycle 3 |  | 4.2 (4.0)
  Overall Responders and Non-Responders - Cycle 4: number analyzed (Participants) | 4 | 0
  Overall Responders and Non-Responders - Cycle 4 | 3.2 (2.0) |
  Overall Responders and Non-Responders - Cycle 5: number analyzed (Participants) | 0 | 1
  Overall Responders and Non-Responders - Cycle 5 |  | 0.2
  Overall Responders and Non-Responders - Cycle 6: number analyzed (Participants) | 2 | 0
  Overall Responders and Non-Responders - Cycle 6 | 2.7 (0.9) |

5. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 20 months and 18 days for the first Arm/Group, and 28 months and 23 days for the second Arm/Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Glioblastoma or Gliosarcoma With No Prior Bevacizumab Exposure | Glioblastoma or Gliosarcoma With Prior Bevacizumab Exposure
Number analyzed (Participants) | 9 | 26
Participants | 9 | 21

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 20 months and 18 days for the first Arm/Group, and 28 months and 23 days for the second Arm/Group.
Arm/Group | Glioblastoma or Gliosarcoma With No Prior Bevacizumab Exposure | Glioblastoma or Gliosarcoma With Prior Bevacizumab Exposure
All-Cause Mortality (participants affected / at risk) | 9/9 | 20/26
Serious Adverse Events (participants affected / at risk) | 2/9 | 7/26
Other Adverse Events (participants affected / at risk) | 9/9 | 21/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glioblastoma or Gliosarcoma With No Prior Bevacizumab Exposure (N=9) | Glioblastoma or Gliosarcoma With Prior Bevacizumab Exposure (N=26)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glioblastoma or Gliosarcoma With No Prior Bevacizumab Exposure (N=9) | Glioblastoma or Gliosarcoma With Prior Bevacizumab Exposure (N=26)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Alanine aminotransferase increased (Investigations) | 1 (2) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, Blood in stool (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, Elevated ALT (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Blood and lymphatic system disorders - Other, Elevated AST (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 3 (3)
Bronchial infection (Infections and infestations) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 3 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 8 (9)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Eye disorders - Other, Right Hemianops (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Left upper quadrant defect (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fatigue (General disorders) | 6 (6) | 12 (13)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 2 (2) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Intermittent blood in stool (Hematochezia) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Mouth sores (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Sphincter Dysfunction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (5) | 6 (7)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 7 (22) | 11 (27)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Investigations - Other, Abnormal taste (Investigations) | 0 (0) | 1 (1)
Investigations - Other, Elevated TSH (Investigations) | 0 (0) | 1 (1)
Investigations - Other, Hemiparesis (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 3 (3)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 8 (11)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — - Other, GBM (Extraocular movements, confusion)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) — - Other, Numbness/tingling, right sided weakness, & headaches
Nervous system disorders - Other, Skin sensitivity to touch (Nervous system disorders) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 2 (5) | 3 (5)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 4 (4)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Runny nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 3 (3) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Lacerations on legs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (6) | 0
Skin and subcutaneous tissue disorders - Other, Cushingoid facies-right cheek (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Spasticity (Nervous system disorders) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (8)
Weight loss (Investigations) | 2 (2) | 3 (3)
White blood cell decreased (Investigations) | 3 (8) | 1 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT01931098/Prot_SAP_001.pdf
  • Informed Consent Form (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT01931098/ICF_002.pdf